CLINICAL TRIAL: NCT04301635
Title: Upper-airway Changes After Bimaxillary Advancement in Moderate-severe Obstructive Sleep Apnoea / Hypopnoea Syndrome
Brief Title: Upper-airway Changes After Bimaxillary Advancement in OSAHS
Acronym: OSAHS
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital de Cruces (Other)
Collaborators: University of the Basque Country (UPV/EHU) (Other); Biobizkaia Health Research Institute (Other Government)
Responsible Party: Principal Investigator, Carlos Prol Teijeiro, Oral & Maxillofacial Consultant, Hospital de Cruces
Other Study IDs: SAHS_PROL
Record Dates: First submitted 2020-03-04; First posted 2020-03-10 (Actual); Last update posted 2021-02-10 (Actual); Status verified 2021-02

CONDITIONS: OSAHS; Craniofacial Abnormalities
Keywords: OSAHS; Sleep disorder; Orthognathic surgery; Maxillomandibular advancement; Counterclockwise rotation
MeSH Terms: conditions — Sleep Apnea, Obstructive; Craniofacial Abnormalities; Sleep Wake Disorders | interventions — Orthognathic Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preoperative (Pre-): Moderate-severe obstructive sleep apnoea / hypopnoea patients, preoperative
  Interventions: Procedure: Maxillo-mandibular Advancement + Counterclockwise rotation
- Postoperative (Post-): Moderate-severe obstructive sleep apnoea / hypopnoea patients, postoperative
  Interventions: Procedure: Maxillo-mandibular Advancement + Counterclockwise rotation

INTERVENTIONS:
Procedure: Maxillo-mandibular Advancement + Counterclockwise rotation — Maxilla: Lefort I osteotomy Mandible: Obwegeser-Dal-Pont osteotomy Movements: Advance and counterclockwise rotation
  Other Names: Bimaxillary Advancement; Orthognathic Surgery

SUMMARY:
One of the most effective surgical treatments for obstructive sleep apnoea / hypopnoea syndrome (SAHS) with global impact on the upper-airway (UA) is the maxilla-mandibular advancement (MMA). Retrospective-prospective observational study of: clinical outcomes, UA and dental-cranium-facial (DCF) morphology.

Population sample will be patients treated in the Maxillofacial Surgery department of "Hospital de Cruces". As inclusion criteria: ≥18 years-old, moderate-severe SAHS in supine position, multidisciplinary committee of sleep pathology evaluation for surgical indication, and written informed consents. As exclusion criteria: pregnant woman, SAHS of central origin, cranium-facial deformities that significantly modify normal UA, different surgery than MMA and inconclusive / incomplete tests. It is estimated ≥90% males; ≥90% 30-59 years-old; ≤10% extreme weights; 25% complementary surgeries; and sample size 40. Medical ethics code of the Declaration of Helsinki will be taken into account. To collect the pre- / postoperative data we will use, calibrated and standardized: polysomnography (PSG), computed tomography (CT), right face profile picture (RFP) and lateral teleradiography of the cranium (LTC). Furthermore, the Epworth scale and non-validated subjective self-perception test of facial aesthetics will be performed.

Clinical outcomes will be evaluated from PSG using apnoea / hypopnoea index and pulse oximeter oxygen saturation, and from Epworth scale. UA morphology from CT, globally and by specific locations, through lengths, volumes, areas, dimensions, and other measurements. DCF aspects from RFP and LTC, by Ricketts cephalometric basic analysis and facial aesthetics test. Statistical, descriptive analysis of frequencies and comparative by pairs of quantitative data will be by t-Student or Wilcoxon test, after checking the variables normality with the Kolmogorov-Smirnov test.

DETAILED DESCRIPTION:
HYPOTHESIS:

H0: Upper-airway (UA) morphology does not change as a consequence of maxilla-mandibular advancement (MMA) in patients with moderate-severe obstructive sleep apnoea / hypopnoea syndrome (SAHS).

H1: UA changes as a consequence of MMA in patients with moderate-severe SAHS. To answer this hypothesis, the following will be determined: Vertical UA length, volume, axial areas, ellipticity, uniformity, prevertebral soft tissue (PST) and soft palate (SP) lengths and position of the hyoid bone.

As secondary hypotheses:

H0: Clinical outcomes of MMA in moderate-severe SAHS are not successful. H1: Clinical outcomes of MMA in moderate-severe SAHS are successful. To answer, the apnoea / hypopnoea index (AHI), pulse oximeter oxygen saturation (SPO2) and daytime sleepiness will be determined.

H0: DCF morphology is unfavourable as a result of MMA in moderate-severe SAHS. H1: DCF morphology is not unfavourable as a result of MMA in moderate-severe SAHS.

To answer, the parameters of the Ricketts cephalometric basic analysis will be quantified and interpreted, and the patient's self-perception will be assessed.

OBJECTIVES:

Specify and quantify morphological changes in key anatomical locations of the UA by computed tomography (CT), in terms of vertical lengths, volumes, areas, axial dimensions, and other measurements. These changes happen after MMA surgery in patients diagnosed with moderate-severe SAHS from a representative cohort. We are intended to demonstrate: shortening, increase in volume and areas, more elliptical and uniform shape, modifications of PST and SP and more anterior-superior hyoid bone position.

As secondary objectives, inherent to the treatment received, it is first intended to determine and evaluate clinical outcomes: objectively by polysomnography, and subjectively by the Epworth scale. Secondary, it is intended to specify and quantify changes in DCF morphology: objectively by a two-dimensional cephalometric analysis from lateral teleradiography of the cranium (LTC) and right face profile picture (RFP), and subjectively by a non-validated facial aesthetics test (FAT).

DESIGN:

Observational retrospective-prospective study, which does not make any modification of the usual clinical practice (surgical indication criteria, procedures, examinations, surgical techniques...), of: clinical outcomes, UA morphology, and DCF aspects of SAHS patients undergoing MMA.

* Logistic and organizational process for the participants: Explanations, invitation to participate, resolution of doubts, delivery of written information sheet and informed consent, collection of them and FAT. Everything will be done in two face-to-face clinic consultations that are already part of the usual work protocol of the Maxillofacial Surgery department of our hospital for patients with SAHS. It is estimated that it only involves about 10-15 minutes per consultation of extra time, without the need of additional specific appointments for the present study. With regard to clinical history, complementary examinations and surgical procedure, nothing additional is required regarding the usual workflow for SAHS patients in our department.
* Logistic and organizational process for researchers: It is based on office and digital work, without biological samples.

A sample size of 40 subjects is estimated, compiling previous studies and the Granmo® calculator. This would achieve significant statistics in all the parameters considered to answer the main hypothesis, and most of the secondary ones.

The Declaration of Helsinki code of medical ethics for research in human beings will be taken into account, protecting the health of the participant, being voluntary the inclusion, interrupting the investigation if it can be detrimental to the well-being of the participant and agreement of confidentiality in the IC. The "CEIC OSI Exkerraldea-Enkarterri-Cruces" committee has approved the study (Code CEIC E19/39).

DATA ANALYSIS:

We will analyze the qualitative and continuous quantitative variables in categorical variables. Descriptive statistics of frequencies will be calculated. For statistical inference, only comparisons are made between two continuous variables, all dependent and paired (pre- / post-). To verify that the variables follow a normal distribution, the Kolmogorov-Smirnov statistic will be used. The comparisons will then be made with the t-Student test for two dependent samples or the Wilcoxon ranks test if they do not follow a normal distribution. Statistically significant results will be considered if p ˂0.05.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years-old.
* Diagnosis by polysomnography of moderate-severe obstructive sleep apnoea / hypopnoea syndrome (SAHS) in supine position.
* Approval of the surgical indication by the multidisciplinary sleep committee of our hospital
* Written informed consent (IC) of photography or image recording, orthognathic surgery program inclusion and facial deformity surgery.
* Specific IC for inclusion in the present study.

Exclusion Criteria:

* Pregnant woman
* Central SAHS
* Medical-surgical history that significantly alter the normal upper-airway anatomy: trauma, tumour, major congenital craniofacial deformity
* Different orthognathic surgery than MMA
* Inconclusive / incomplete tests and data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients treated in a single centre: Maxillofacial Surgery department, "Hospital de Cruces", Barakaldo, Spain Time period from 01/01/2012 to 01/31/2019.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2019-02-04 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Upper-airway morphology: Vertical length | Through study completion, an average of 1 year
  From computed-tomography examinations. Total, retropalatal compartment, retro-glossal compartment, hypopharynx compartment and summatory. Measured in mm.
Upper-airway morphology: volume | Through study completion, an average of 1 year
  From computed-tomography examinations. Total, retropalatal compartment, retro-glossal compartment, hypopharynx compartment and summatory. Measured in mm^3.
Upper-airway morphology: area | Through study completion, an average of 1 year
  From computed-tomography examinations. Minimum, hard palate plane, parallel uvula tip plane, parallel epiglottis tip plane, parallel inferior edge of the hyoid bone plane. Measured in mm. Measured in mm^2.
Upper-airway morphology: ellipticity | Through study completion, an average of 1 year
  A formula: transversal dimension / anteroposterior dimension. Dimensions characteristics are: From computed-tomography examinations. Minimum, hard palate plane, parallel uvula tip plane, parallel epiglottis tip plane, parallel inferior edge of the hyoid bone plane. Measured in mm.
Upper-airway morphology: uniformity | Through study completion, an average of 1 year
  A formula: minimum area / (hard palate area + uvula tip area + epiglottis tip area + hyoid bone area) Measured in units from 0 to 1.
Upper-airway morphology: prevertebral soft tissue length | Through study completion, an average of 1 year
  From computed-tomography examinations. Measured in mm.
Upper-airway morphology: soft palate length | Through study completion, an average of 1 year
  From computed-tomography examinations. Measured in mm.
Upper-airway morphology: position of the hyoid bone | Through study completion, an average of 1 year
  From computed-tomography examinations. Measured in mm in the anteroposterior aspect and also the superoinferior aspect, this one is the same measure as vertical length.

SECONDARY OUTCOMES:
Clinical outcomes: Apnoea / hypopnoea index | Through study completion, an average of 1 year
  From polysomnography records. Global, in supine position and in lateral position. Measured in units from 0 to 100.
Clinical outcomes: pulse oximeter oxygen saturation. | Through study completion, an average of 1 year
  From polysomnography records. Mean, basal and minimum. Measured in %.
Clinical outcomes: daytime sleepiness | Through study completion, an average of 1 year
  From the Epworth scale. Measured in units from 0 to 24.
Dental-cranium-facial morphology: Ricketts cephalometric basic analysis: facial axis angle | Through study completion, an average of 1 year
  From lateral teleradiography of the cranium and right facial profile photography. Measured in grades.
Dental-cranium-facial morphology: Ricketts cephalometric basic analysis: facial depth | Through study completion, an average of 1 year
  From lateral teleradiography of the cranium and right facial profile photography. Measured in grades.
Dental-cranium-facial morphology: Ricketts cephalometric basic analysis: mandibular plane angle | Through study completion, an average of 1 year
  From lateral teleradiography of the cranium and right facial profile photography. Measured in grades.
Dental-cranium-facial morphology: Ricketts cephalometric basic analysis: lower facial height | Through study completion, an average of 1 year
  From lateral teleradiography of the cranium and right facial profile photography. Measured in mm.
Dental-cranium-facial morphology: Ricketts cephalometric basic analysis: mandibular arch | Through study completion, an average of 1 year
  From lateral teleradiography of the cranium and right facial profile photography. Measured in grades.
Dental-cranium-facial morphology: Ricketts cephalometric basic analysis: facial convexity | Through study completion, an average of 1 year
  From lateral teleradiography of the cranium and right facial profile photography. Measured in mm.
Dental-cranium-facial morphology: Ricketts cephalometric basic analysis: maxillary depth | Through study completion, an average of 1 year
  From lateral teleradiography of the cranium and right facial profile photography. Measured in grades
Dental-cranium-facial morphology: Ricketts cephalometric basic analysis: incisor protrusion | Through study completion, an average of 1 year
  From lateral teleradiography of the cranium and right facial profile photography. Measured in mm.
Dental-cranium-facial morphology: Ricketts cephalometric basic analysis: incisor inclination | Through study completion, an average of 1 year
  From lateral teleradiography of the cranium and right facial profile photography. Measured in grades.
Dental-cranium-facial morphology: Ricketts cephalometric basic analysis: incisor extrusion | Through study completion, an average of 1 year
  From lateral teleradiography of the cranium and right facial profile photography. Measured in mm.
Dental-cranium-facial morphology: Ricketts cephalometric basic analysis: interincisal angle | Through study completion, an average of 1 year
  From lateral teleradiography of the cranium and right facial profile photography. Measured in grades.
Dental-cranium-facial morphology: Ricketts cephalometric basic analysis: upper molar position | Through study completion, an average of 1 year
  From lateral teleradiography of the cranium and right facial profile photography. Measured in mm.
Dental-cranium-facial morphology: Ricketts cephalometric basic analysis: labial protrusion | Through study completion, an average of 1 year
  From lateral teleradiography of the cranium and right facial profile photography. Measured in mm.
Dental-cranium-facial morphology: non-validated facial aesthetics test: general satisfaction | Through study completion, an average of 1 year
  Qualitative measurement: none, little, ok, a lot of.
Dental-cranium-facial morphology: non-validated facial aesthetics test: modifications perceived by the patient | Through study completion, an average of 1 year
  Qualitative measurement: much worse, worse, no changes, better, much better.
Dental-cranium-facial morphology: non-validated facial aesthetics test: modifications perceived by family members and friends | Through study completion, an average of 1 year
  Qualitative measurement: much worse, worse, no changes, better, much better.
Dental-cranium-facial morphology: non-validated facial aesthetics test: smile | Through study completion, an average of 1 year
  Qualitative measurement: much worse, worse, no changes, better, much better.
Dental-cranium-facial morphology: non-validated facial aesthetics test: face rejuvenation | Through study completion, an average of 1 year
  Qualitative measurement: older, no changes, younger.
Dental-cranium-facial morphology: non-validated facial aesthetics test: face slimness | Through study completion, an average of 1 year
  Qualitative measurement: bulkier, no changes, slimmer.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Prol, Mr, Principal Investigator — Osakidetza
Locations (1):
- Carlos Prol, Barakaldo, Bizkaia, Spain

IPD SHARING:
Plan to Share IPD: Undecided
General non-identifying subjects data Upper-airway morphology data Clinical outcomes data Dental-cranium-facial morphology data